CLINICAL TRIAL: NCT01742182
Title: Circadian Rhythms and Sleep-Wake Cycles in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Aleksandar Videnovic, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Circadian Rhythms in PD; 1K23NS072283-01A1 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Excessive Daytime Sleepiness; Circadian Rhythms; Light Therapy
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention)
- PD patients without sleep problems (No Intervention)
- PD patients with sleep problems (Active Comparator): light exposure
  Interventions: Other: Light exposure
- PD patients with sleep problem (Placebo Comparator): light exposure
  Interventions: Other: Light exposure

INTERVENTIONS:
Other: Light exposure
  Arms: PD patients with sleep problem; PD patients with sleep problems

SUMMARY:
Disruption of sleep and alertness is one of the most disabling non-motor symptoms of Parkinson's disease (PD). Mechanisms leading to impaired sleep and alertness in PD are not well understood, and treatment options remain limited. The proposed research will examine markers of the circadian system, sleepiness and sleep quality in PD patients and healthy controls. Further, the project will examine effects of bright light exposure on circadin function, sleep and alertness in PD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD as defined by the United Kingdom PD Society Brain Bank Criteria;
2. PD Hoehn and Yahr stage 2-4;
3. Pittsburgh Sleep Quality Index (PSQI) score >5 in group 1, and ≤5 in group 2;
4. Epworth Sleepiness Scale (ESS) score ≥10 in group 1, and <10 in group 2;

Control participants will be matched for gender and age with PD participants.

Exclusion Criteria:

1. Atypical or secondary forms of Parkinsonism;
2. Cognitive impairment as determined by the Mini-Mental State Examination (MMSE) score of ≤ 26;
3. Presence of depression defined as the Beck Depression Inventory (BDI) score >14;
4. Use of hypno-sedative drugs for sleep or stimulants; participants will be allowed to taper these drugs and will become eligible at least 4 weeks after the taper is completed;
5. Use of SSRIs / SNRIs antidepressants, unless the participant has been on a stable dose for at least 3 months prior to the screening;
6. Use of medications known to affect melatonin secretion;
7. Unstable/serious medical illness.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
circadian rhythm of melatonin | June 2012- May 2017
Sleep Efficiency | June 2012- May 2017
Daytime Somnolence | June 2012- May 2017

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Videnovic, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States